CLINICAL TRIAL: NCT04618575
Title: A Randomized Controlled Open-label Clinical Trial of Ursodeoxycholic Acid Combined With Total Glucosides of Paeony in the Treatment of PBC With AIH Features 1
Brief Title: Ursodeoxycholic Acid Combined With Total Glucosides of Paeony in the Treatment of PBC With AIH Features 1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC with AIH features 1
Record Dates: First submitted 2020-10-31; First posted 2020-11-06 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis; Primary Biliary Cholangitis; Autoimmune
MeSH Terms: conditions — Hepatitis; Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursodeoxycholic acid combined with total glucosides of paeony (Experimental)
  Interventions: Drug: Ursodeoxycholic acid combined with total glucosides of paeony
- Ursodeoxycholic acid only (Other)
  Interventions: Drug: Ursodeoxycholic acid only

INTERVENTIONS:
Drug: Ursodeoxycholic acid combined with total glucosides of paeony — Ursodeoxycholic acid combined with total glucosides of paeony
  Arms: Ursodeoxycholic acid combined with total glucosides of paeony
Drug: Ursodeoxycholic acid only — Ursodeoxycholic acid only
  Arms: Ursodeoxycholic acid only

SUMMARY:
A randomized controlled open-label clinical trial of ursodeoxycholic acid combined with total glucosides of paeony in the treatment of PBC with AIH features 1

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years;
2. The diagnosis of PBC is clear and does not meet the Paris criteria for diagnosing PBC overlap AIH, but it needs to meet 1.0xULN < ALT ≤ 3.0xULN or 1.0xULN < AST ≤ 3.0xULN or 1.0xULN < IgG ≤ 1.3xULN, and liver pathological biopsy excludes moderate or higher interface inflammation;
3. Agreed to participate in the trial, and assigned informed consent.

Exclusion Criteria:

1. The presence of hepatitis A, B, C, D, or E virus infection;
2. Patients with presence of cirrhosis;
3. Patients with presence of fulminant liver failure;
4. Liver damage caused by other reasons: such as primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson's disease;
5. Pregnant and breeding women and women of childbearing age in need of reproduction;
6. Severe disorders of other vital organs, such as severe heart failure, cancer;
7. Parenteral administration of blood or blood products within 6 months before screening;
8. Recent treatment with drugs having known liver toxicity;
9. Taken part in other clinic trials within 6 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-11-05 (Estimated); Study Completion 2022-11-05 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission | up to 12 months
  The percentage of patients in biochemical remission, defined as normalization of serum ALT and IgG levels after 24 weeks of treatment, per treatment group.

SECONDARY OUTCOMES:
Partial remission | up to 12 months
  Partial remission, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) serum levels >1x Upper Limit of Normal (ULN) and <2x ULN
Minimal response | up to 12 months
  Minimal response, defined as decrease of ALT or AST serum levels but still >2x ULN
Treatment failure | up to 12 months
  defined as no improvement or increase of ALT or AST serum levels
Side-effects | up to 12 months
  Drug related side-effects
Clinical symptoms | up to 12 months
  Jaundice, fatigue, itching, etc
Changes in the proportion of blood immune cells | up to 12 months
  percentage of T cells, DC, MDSC, Treg, Breg, plasma cells, NK, NKT

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No